CLINICAL TRIAL: NCT00654017
Title: Multicenter, Double-Blind, Randomized, Placebo-controlled Study of Flexible, Titration Dose Administered on an As Needed Basis (PRN) to Evaluate the Efficacy and the Safety of Sildenafil for the Treatment of Erectile Dysfunction in Male Patients on Hemodialysis
Brief Title: A Study Evaluating the Efficacy and Safety of Sildenafil in Patients With Erectile Dysfunction Receiving Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481076
Record Dates: First submitted 2008-03-31; First posted 2008-04-07 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Disfunction; Hemodialysis
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- sildenafil (Active Comparator)
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: placebo — Placebo comparator to be given per protocol.
  Arms: placebo
Drug: sildenafil — oral sildenafil citrate at an initial dose of 25 mg, which could have been up-titrated to 50 mg at Visit 3 based on the patient's efficacy, safety and tolerability responses; at Visits 4 and 5, the dose could remain the same, be increased to 100 mg, or decreased to 25 mg depending on the safety, efficacy, and tolerability
  Arms: sildenafil

SUMMARY:
The study was done to evaluate the efficacy, safety, and tolerability of orally administered sildenafil taken as needed about one hour before sexual activity after a 10-week period in male outpatients with erectile dysfunction and severe renal failure who were on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Included patients had been in a stable relationship with a female partner for at least 6 months
* A diagnosis of renal failure, with creatinine clearance ≤10 ml/min; been under hemodialysis for at least 6 months prior to the screening period, and a clinical diagnosis of erectile dysfunction (ED) as confirmed by International Index of Erectile Function (IIEF-5) score of <21 and defined as an "incapacity to obtain and/or maintain an erection sufficient for a satisfactory sexual performance".

Exclusion Criteria:

* Patients in regular use of nitrates or nitric oxide donor drugs, or have received a prescription to use these substances in any formulation
* Patients with genital anatomic malformation that may significantly impair erection (e.g., serious penile fibrosis)
* Patients with other sexual disorders (e.g., hypoactive sexual desire) considered as a primary diagnosis, with a coexisting ED diagnosis, including patients receiving anti-androgenic therapy whose libido has not been preserved; patients receiving hormonal replacement therapy for at least 6 months, or whose dose has not been stabilized within the last 6 months before the study screening period
* Patients with diabetes mellitus presenting poor control of their diabetes and/or proliferate diabetes retinopathy.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-10; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Response to questions 3 (frequency of penetration) and 4 (frequency of maintained erection) of the International Index of Erectile Function (IIEF). | Baseline and Week 10

SECONDARY OUTCOMES:
rate of successful sexual intercourse (number of attempts at sexual intercourse, number of successful attempts and percentage of attempts that were successful) | Baseline to Week 10
response to Partner's Satisfaction Questionnaire (optional) | Week 10
total Score of Quality of Life and erectile dysfunction questionnaire | Baseline and Week 10
monitoring of adverse events (AEs) and measurement of sitting blood pressure and heart rate | Baseline, and Weeks 2, 4, 6, and 10
response to Question 1 of the Global Efficacy Assessment Question | Week 10
responses to questions of the IIEF | Baseline and Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Brazil (7):
  - Pfizer Investigational Site, Fortaleza, Ceará
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Londrina, Paraná
  - Pfizer Investigational Site, Jaú, São Paulo
  - Pfizer Investigational Site, São José do Rio Preto, São Paulo
  - Pfizer Investigational Site, Sorocaba, São Paulo
  - Pfizer Investigational Site, São Paulo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481076&StudyName=A%20Study%20Evaluating%20the%20Efficacy%20and%20Safety%20of%20Sildenafil%20for%20the%20Treatment%20of%20Erectile%20Dysfunction%20in%20Male%20Patients%20on%20Hemodialysis.